CLINICAL TRIAL: NCT05174832
Title: Induction of Cisplatin/Nab-paclitaxel/Pembrolizumab Followed by Olaparib/Pembrolizumab Maintenance in Triple-negative Metastatic Breast Cancer Patients
Brief Title: Induction of Cisplatin/Nab-paclitaxel/Pembrolizumab Followed by Olaparib/Pembrolizumab Maintenance in mTNBC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Xichun Hu, M.D. , ph.D., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMPLEMENT
Record Dates: First submitted 2021-12-13; First posted 2022-01-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-11

CONDITIONS: Triple Negative Breast Cancer
Keywords: Pembrolizumab; Olaparib; Platinum-based chemotherapy; Triple negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Cisplatin; 130-nm albumin-bound paclitaxel; pembrolizumab; olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cisplatin+ Nab-paclitaxel + Pembrolizumab followed by Pembrolizumab monotherapy (Active Comparator): 4~6 cycles combination therapy of Cisplatin, Nab-paclitaxel and Pembrolizumab as induction therapy; Pembrolizumab monotherapy as maintenance therapy
  Interventions: Drug: Cisplatin; Drug: Nab-paclitaxel; Drug: Pembrolizumab
- Cisplatin+Nab-paclitaxel+Pembrolizumab followed by Pembrolizumab+Olaparib (Experimental): 4~6 cycles combination therapy of Cisplatin, Nab-paclitaxel and Pembrolizumab as induction therapy; Pembrolizumab plus Olaparib as maintenance therapy
  Interventions: Drug: Cisplatin; Drug: Nab-paclitaxel; Drug: Pembrolizumab; Drug: Olaparib

INTERVENTIONS:
Drug: Cisplatin — 75 mg/m2 IV days 1 of each 21-day cycle
Drug: Nab-paclitaxel — 125 mg/m2 IV days 1 and 8 of each 21-day cycle
Drug: Pembrolizumab — 200 mg IV every 21 days
  Other Names: keytruda
Drug: Olaparib — 300 mg PO BID
  Other Names: LYNPARZA
  Arms: Cisplatin+Nab-paclitaxel+Pembrolizumab followed by Pembrolizumab+Olaparib

SUMMARY:
This study aims to investigate if olaparib plus pembrolizumab will maintain the clinical benefit achieved after induction therapy with Albumin-bound paclitaxel combined with cisplatin(AP) regimen and pembrolizumab in previously untreated locally advanced, recurrent or metastatic TNBC population with PD-L1 CPS≥1.

DETAILED DESCRIPTION:
TNBC is a hard-to-treat disease requiring continuous administration of drugs, necessitating further exploration of optimal maintenance strategy. However, there are currently no standard maintenance treatment regimens in the treatment of mTNBC. KEYNOTE-355 has already proved pembrolizumab has durable antitumor activity and manageable safety in patients with metastatic TNBC. Olaparib is now established as maintenance therapy for platinum-sensitive populations regardless of BRCA status in the setting of other tumor types. Furthermore, preclinical and clinical data indicates that olaparib and pembrolizumab combination have an improved therapeutic effect, showing promising synergistic benefits. Therefore, adding olaparib to pembrolizumab after induction treatment with a platinum-based regimen plus pembrolizumab will high likely change and expand the treatment paradigm in this disease, particularly for those patients with platinum-sensitive TNBC tumors. Olaparib plus pembrolizumab has the potential for further treatment benefit as a chemo-sparing regimen.

ELIGIBILITY:
Inclusion Criteria:

Induction period:

* Locally advanced, recurrent or metastatic TNBC that has not been treated with chemotherapy for the advanced disease. Local or distant disease recurrence must be≥6 months from the completion of the last dose of chemotherapy.
* PD-L1 CPS≥1 and ER and PR negative, HER2 negative breast cancer.
* Archival tumor tissue sample or newly obtained core or excisional biopsy sample
* Measurable disease based on RECIST 1.1.
* ECOG Performance Status 0-1
* Life expectancy≥18 weeks
* Adequate hematological, renal and hepatic function according to all of the following laboratory values (to be performed within 10 days prior to start of study treatment)

Maintenance period：

* Complete induction therapy without permanent discontinuation of pembrolizumab, nab-paclitaxel or cisplatin.
* CR, PR, or SD status based on RECIST 1.1 as determined by local investigators.
* ECOG Performance Status 0-1, as assessed within 7 days prior to the start of maintenance therapy.
* Recovery of toxicities related to induction therapy to ≤ grade 1 (except alopecia) prior to randomization. Grade 2 neuropathy will be allowed, whereas grade 2 hyperthyroidism or hypothyroidism will also be allowed if it can be well controlled with medicines.

Exclusion Criteria:

Induction period:

* Has received any prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Has received any prior therapy with either olaparib or other PARP inhibitors.
* Has received any prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.
* Has received prior radiotherapy within 2 weeks of start of study treatment
* Has received a live vaccine within 30 days prior to the first dose of study drug
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, cervical cancer in situ) that have undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a known history of hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipient
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has gastrointestinal impairment that could affect their ability to take or absorb oral medicines; evidence of severe or uncontrolled cardiac disease; active bleeding or bleeding diathesis defined as significant hemorrhage; or hemoptysis.
* Has a resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions or has congenital long QT syndrome.
* Has myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or has features suggestive of MDS/AML
* Has a history of (non-infectious) pneumonitis that required treatment with steroids; or current pneumonitis.
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of active Hepatitis B or known active Hepatitis C virus infection
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Has been pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.
* Failure to comply with the study procedures, restrictions and requirements of the study

Maintenance period：

* Has permanently discontinued from nab-paclitaxel, cisplatin or pembrolizumab during induction period due to toxicity.
* Currently receiving either strong or moderated inhibitors of cytochrome P450 (CYP) 3A4 that cannot be discontinued for the duration of the study.
* Currently receiving either strong or moderate inducers of CYP3A4 that cannot be discontinued for the duration of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by local investigators | Up to 36 months
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by investigators | Up to 36 months
  PFS is defined as the time from enrollment data (informed consent date) to the first documented disease or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 36 months
  OS is defined as the time from enrollment date to death due to any cause.
Objective Response Rate(ORR) in induction and maintenance phase | Up to approximately 36 months
  ORR is defined as the proportion of the total number of subjects with a confirmed CR or confirmed PR
Progression-Free Survival (PFS) in gBRCAm and gBRCAwt participants | Up to approximately 36 months
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first.
Overall Survival (OS) in gBRCAm and gBRCAwt participants | Up to approximately 36 months
  OS: the time from randomization to death due to any cause.
Progression-Free Survival (PFS) in HRR deficient participants | Up to approximately 36 months
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first.
Overall Survival (OS) in HRR deficient participants | Up to approximately 36 months
  OS: the time from randomization to death due to any cause.
Overall Survival (OS) | Up to approximately 36 months
  OS: the time from randomization to death due to any cause.
Number of Participants with Treatment Related Adverse Events | Up to approximately 36 months
  AEs assessed by CTCAE V5.0

OTHER OUTCOMES:
Molecular biomarkers that might be indicative of clinical response/resistance | Up to approximately 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China